CLINICAL TRIAL: NCT06793072
Title: Assessment of Adipokine Concentrations and Their Association With the Metabolic Profile of Women With PCOS
Brief Title: Adipokines in Polycystic Ovary Syndrome
Status: Recruiting | Type: Observational
Sponsor: Jagiellonian University (Other)
Responsible Party: Principal Investigator, Iwona Magdalena Gawron, PhD, MD, Principal Investigator, Jagiellonian University
Other Study IDs: 1072.6120.44.2024
Record Dates: First submitted 2025-01-20; First posted 2025-01-27 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: PCOS; Reproductive Age
Keywords: insulin resistance; polycystic ovary syndrome; metabolic syndrome; adipokines
MeSH Terms: conditions — Insulin Resistance; Polycystic Ovary Syndrome; Metabolic Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood serum
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- PCOS+IR: Polycystic ovary syndrome + insulin resistance
  Interventions: Diagnostic Test: Leptin concentration in blood serum; Diagnostic Test: Resistin concentration in blood serum; Diagnostic Test: Omentin-1 concentration in blood serum
- PCOS + no IR: Polycystic ovary syndrome + no insulin resistance
  Interventions: Diagnostic Test: Leptin concentration in blood serum; Diagnostic Test: Resistin concentration in blood serum; Diagnostic Test: Omentin-1 concentration in blood serum
- No PCOS: Women without PCOS (control)
  Interventions: Diagnostic Test: Leptin concentration in blood serum; Diagnostic Test: Resistin concentration in blood serum; Diagnostic Test: Omentin-1 concentration in blood serum

INTERVENTIONS:
Diagnostic Test: Leptin concentration in blood serum — Fasting plasma leptin concentration measurement with results expressed in pg/ml and comparison across all study arms
Diagnostic Test: Resistin concentration in blood serum — Fasting plasma resistin concentration measurement with results expressed in pg/ml and comparison across all study arms
Diagnostic Test: Omentin-1 concentration in blood serum — Fasting plasma omentin-1 concentration measurement with results expressed in pg/ml and comparison across all study arms

SUMMARY:
The aim of the study is to compare the concentrations of leptin, resistin, and omentin-1 in women across three research groups: those with polycystic ovary syndrome without insulin resistance, those with polycystic ovary syndrome with insulin resistance, and women without polycystic ovary syndrome.

DETAILED DESCRIPTION:
Polycystic ovary syndrome (PCOS) is the most prevalent endocrinopathy among reproductive-age women, characterized primarily by insulin resistance (IR), which has a prevalence of 35% to 80%. Metabolic disturbances associated with PCOS contribute to a higher incidence of cardiovascular diseases and endometrial cancer prior to menopause. The hyperinsulinemic-euglycemic clamp study is regarded as the gold standard for assessing insulin sensitivity; however, its clinical application is limited. Alternative assessments, such as the Homeostasis Model Assessment of Insulin Resistance (HOMA-IR) and fasting insulin or glucose tolerance tests, provide limited clinical utility. Therefore, there is a pressing need for the identification of more precise and universal markers of insulin resistance. There is a need to elucidate the precise role of adipokines in the etiology of PCOS and their association with insulin resistance, which is responsible for the development of adverse health-related complications.

The aim of the study is to measure and compare the concentrations of selected adipokines: leptin, resistin, omentin-1 across three research groups: those with polycystic ovary syndrome without insulin resistance, those with polycystic ovary syndrome with insulin resistance, and women without polycystic ovary syndrome.

The tests will be performed using immunoenzymatic methods (ELISA) and the Erba XL biochemical analyzer.

The concentrations of the investigated substances will be measured and compared within the three research groups.

Statistical analysis will be conducted using SPSS Statistics software.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-45

Exclusion Criteria:

* previous removal of at least one ovary
* treated diabetes of any type
* diagnosed and treated metabolic diseases
* diagnosed and treated autoimmune diseases
* diagnosed and treated autoinflammatory diseases(Edited)Restore original

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: women aged 18-45 years managed for menstrual irregularities or routine check-up
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-01-20 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Comparison of resistin concentration in three study groups | up to 6 months
  Measurement and comparison of mean fasting plasma resistin concentration expressed in pg/ml in three study groups
Comparison of leptin concentration three study groups | up to 6 months
  Measurement and comparison of mean fasting plasma leptin concentration expressed in pg/ml in three study groups
Comparison of omentin-1 concentration in three study groups | up to 6 months
  Measurement and comparison of mean fasting plasma omentin-1 concentration expressed in pg/ml in three study groups

CONTACTS AND LOCATIONS:
Overall Officials: Kazimierz Pityński, Prof., Ph.D., M.D., Study Chair — Jagiellonian University
Locations (1):
- Jagiellonian Univeristy, Krakow, Poland